CLINICAL TRIAL: NCT02323607
Title: Phase I Study of Pacritinib and Chemotherapy in Patients With Acute Myeloid Leukemia and FLT3 Mutations
Brief Title: Pacritinib and Chemotherapy in Treating Patients With Acute Myeloid Leukemia and FLT3 Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bhavana Bhatnagar (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor-Investigator, Bhavana Bhatnagar, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14169; NCI-2014-02436 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Cytarabine; Daunorubicin; Dichlororibofuranosylbenzimidazole; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (pacritinib, cytarabine, daunorubicin hydrochloride) (Experimental): INDUCTION: Patients receive pacritinib PO on days 1-21, cytarabine IV every 24 hours on days 5-11, and daunorubicin hydrochloride IV every 24 hours on days 5-7. Treatment repeats every 28 days for 1-2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pacritinib; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Cohort B (pacritinib, decitabine) (Experimental): INDUCTION: Patients receive pacritinib PO on days 1-21 and decitabine IV every 24 hours on days 5-14. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients achieving CR will proceed with transplant evaluation (if appropriate). Transplant-ineligible patients will receive maintenance courses of pacritinib PO on days 1-21 and decitabine IV over 1 hour daily on days 1-5. Maintenance courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pacritinib; Drug: Decitabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Pacritinib — Given PO
  Other Names: Oral JAK2 Inhibitor SB1518; SB1518
Drug: Cytarabine — Given IV
  Other Names: CHX-3311; U-19920
  Arms: Cohort A (pacritinib, cytarabine, daunorubicin hydrochloride)
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: DNM; DNR; DRB
  Arms: Cohort A (pacritinib, cytarabine, daunorubicin hydrochloride)
Drug: Decitabine — Given IV
  Other Names: 5AZA; DAC
  Arms: Cohort B (pacritinib, decitabine)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of pacritinib when given together with chemotherapy in treating patients with acute myeloid leukemia that have an abnormal change (mutation) in the fms-related tyrosine kinase 3 (FLT3) gene. Pacritinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine, daunorubicin hydrochloride, and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pacritinib and chemotherapy may be a better treatment for acute myeloid leukemia with FLT3 mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of pacritinib in combination with 7+3 or decitabine (respective cohorts are independent of each other) in patients with newly diagnosed or relapsed/refractory acute myeloid leukemia (AML) with FLT3 mutations.

II. To define the specific toxicities, maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of these combinations.

III. To determine the recommended phase 2 dose (RP2D) of these combinations.

SECONDARY OBJECTIVES:

I. To determine the rate and duration of complete remission (CR) +/- hematologic recovery of pacritinib and 7+3 or decitabine in AML.

II. To determine the overall response rate (ORR) and disease free survival at 1 year.

TERTIARY OBJECTIVES:

I. To conduct pharmacokinetic studies of pacritinib in combination with chemotherapy.

II. To determine the impact of pacritinib on the inhibition of Janus kinase 2 (JAK2), FLT3, AXL receptor tyrosine kinase (AXL), signal transducer and activator of transcription 5A (STAT5), spleen tyrosine kinase (Syk).

III. To examine the exosome, cytokine, and chemokine changes of FLT3 down-stream inhibition by pacritinib.

IV. To examine resistance patterns associated with treatment with pacritinib. V. To examine baseline cytogenetic, GTP binding protein overexpressed in skeletal muscle (GEM) signature, and long non-coding (Lnc) ribonucleic acid (RNA) signature and mutational status of the AML tumor cells to better identify subsets of patients with highest likelihood of responding to therapy.

OUTLINE: This is a dose-escalation study of pacritinib. Patients are assigned to 1 of 2 treatment arms.

COHORT A:

INDUCTION: Patients receive pacritinib orally (PO) on days 1-21, cytarabine intravenously (IV) every 24 hours on days 5-11, and daunorubicin hydrochloride IV every 24 hours on days 5-7. Treatment repeats every 28 days for 1-2 courses in the absence of disease progression or unacceptable toxicity.

COHORT B:

INDUCTION: Patients receive pacritinib PO on days 1-21 and decitabine IV every 24 hours on days 5-14. Treatment repeats every 28 days for 2-4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients achieving CR will proceed with transplant evaluation (if appropriate). Transplant-ineligible patients will receive maintenance courses of pacritinib PO on days 1-21 and decitabine IV over 1 hour daily on days 1-5. Maintenance courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML and the presence of FLT3 mutation
* Patients with secondary AML or therapy related disease (t-AML) are eligible
* If the patient has co-morbid medical illness, life expectancy attributed to this must be greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0mg/dL unless due to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Creatinine (Cr) clearance > 50 mL/min by Cockcroft-Gault calculation
* New York Heart Association (NYHA) congestive heart failure (CHF) class II or better
* Cardiac ejection fraction >= 50% for Arm A, >= 40% for Arm B
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Ability to understand and willingness to sign the written informed consent document
* Human immunodeficiency virus (HIV) infection without history of acquired immune deficiency syndrome (AIDS) and sufficiently high cluster of differentiation (CD)4 cells (> 400/mm^3) and low HIV viral loads (< 30,000 copies/ml plasma) not requiring anti-HIV therapy are eligible

Exclusion Criteria:

* Patients with core-binding factor AML (inv[16], t[8;21]) or t(15;17)
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study; treatment with hydroxyurea is permitted during cycle 1 to maintain white blood cell (WBC) < 40,000/uL
* Patients receiving any other investigational agents or patients that have received other investigational agents within 14 days of enrollment
* Patients with active central nervous system (CNS) malignancy
* Major surgery within 2 weeks before day 1
* Uncontrolled active infection; patients with infection requiring parenteral antibiotics are eligible if the infection is controlled
* Patients with significantly diseased or obstructed gastrointestinal tract
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, myocardial infarction within 6 months prior to enrollment, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening has to be documented by the investigator as not medically relevant
* Patients with serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Pregnant women or women who are breastfeeding are excluded from this study; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patients with advanced malignant solid tumors
* Patients who are not able to swallow capsules or tablets
* Patients with baseline corrected QT (QTc) > 500 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
MTD of pacritinib defined as the highest safely tolerated dose where, at most, one patient experiences DLT in 6 evaluable patients, with the next higher dose having at least 2 patients who experience DLT | 28 days
  Assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03. Toxicities will be tabulated by type and grade and displayed in summary form. Further, all adverse event data that are graded as 3, 4, or 5 and classified as either unrelated or unlikely to be related to study treatment will be reviewed for completeness.

SECONDARY OUTCOMES:
Clinical response according to International Working Group criteria | Up to at least 30 days post-treatment
  The degree of response will be summarized within each stratum and at each dose level. ORR will also be presented for those patients treated at the MTD with an exact 95% confidence interval.
Duration of response | Up to at least 30 days post-treatment
  For patients who achieve complete remission, duration of response will be reported.

OTHER OUTCOMES:
Change in FLT3 and JAK2 expression | Baseline to up to at least 30 days post-treatment
  Expression prior to administration of pacritinib and following treatment with pacritinib will be described graphically using boxplots or summary measures (e.g. mean and standard errors). Trends of dose response will be explored within each stratum, as well as whether targets are being "hit" between the strata. Due to data limitations in early clinical trials, analyses will be descriptive in nature.
Change in various genes/microRNA | Baseline to up to at least 30 days post-treatment
  Expression prior to administration of pacritinib and following treatment with pacritinib will be described graphically using boxplots or summary measures (e.g. mean and standard errors). Trends of dose response will be explored within each stratum, as well as whether targets are being "hit" between the strata. Due to data limitations in early clinical trials, analyses will be descriptive in nature.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Bhatnagar, DO, Principal Investigator — Arthur G. James Cancer Hospital and Solove Research Institute at Wexner Medical Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu